CLINICAL TRIAL: NCT05834049
Title: Virtual Parental Presence on Induction of Anesthesia Versus Premedication With Midazolam: A Non-Inferiority Study
Brief Title: Virtual Parental Presence on Induction of Anesthesia vs Premedication With Midazolam
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69571
Record Dates: First submitted 2023-04-11; First posted 2023-04-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Surgery
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Parental Presence on Induction of Anesthesia group (Experimental): Use of Facetime with child and parents during induction
  Interventions: Behavioral: Virtual Parental Presence on Induction of Anesthesia
- Midazolam Group (Experimental): 0.5 mg/kg oral midazolam (max 20 mg) will be given preoperatively.
  Interventions: Behavioral: Midazolam

INTERVENTIONS:
Behavioral: Virtual Parental Presence on Induction of Anesthesia — Apple Inc's FaceTime™ video application will be used when the child is taken to the operating room
  Other Names: VPPIA
  Arms: Virtual Parental Presence on Induction of Anesthesia group
Behavioral: Midazolam — Preoperative midazolam (0.5 mg/kg of oral midazolam with a maximum dose of 20mg) will be given unless medically contraindicated.
  Arms: Midazolam Group

SUMMARY:
This multi-center, prospective, clinical trial targets recruiting children undergoing inhalational induction of anesthesia. The primary objective of this study is to assess the Modified Yale Preoperative Anxiety Scale during induction between children receiving oral midazolam 0.5 mg/kg (max 20 mg) versus virtual parental presence on induction of anesthesia. Patients will be randomized to one of two groups by block randomization.

ELIGIBILITY:
Inclusion Criteria:

* children from ages 4 years to 8 years old undergoing outpatient surgery
* children identified as needing premedication
* ASA physical status I, II or III
* planned inhalational induction
* children presenting from home prior to surgery (not an inpatient)
* English speaking parents and child

Exclusion Criteria:

* children with developmental delay
* children with psychological / emotional disorders
* children with altered mental status
* children in whom midazolam may be medically contraindicated per the discretion of the anesthesia care team
* children with language barrier
* children who are not accompanied by someone able to consent (ie legal guardian)
* children who are inpatient prior to surgery
* children with expected difficult intubation/airway
* children presenting for emergency surgery
* family history or personal history of malignant hyperthermia / risk of MH
* consent not obtained or withdrawal of consent
* children with past history of violent behaviors during induction of anesthesia
* cancellation of surgery
* patients with a diagnosis of COVID-19 or a patient under investigation for COVID-19, including patients being treated with airborne precautions in the operating room
* receipt of any type of medical sedative prior to induction of anesthesia, including (but not limited to) ketamine, and/or dexmedetomidine.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 322 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Anxiety in children | baseline, immediately after the intervention
  We will be using the modified Yale Preoperative Anxiety Scale (mYPAS) which was developed specifically to measure anxiety at anesthesia induction. It looks at activity, facial expression, alertness and arousal, vocalization and interaction with adults. It has a good validity against the State-Trait Anxiety Inventory for Children, as well as good intra and inter-observer reliability. mYPAS contains 5 items (activity, vocalisation, emotional expressivity, state of apparent arousal, and use of parent). The total score ranges from 0 to 22. Higher scores mean higher levels of anxiety.

SECONDARY OUTCOMES:
Induction compliance | immediately during anesthetic induction
  The Induction Compliance Checklist (ICC) is a validated observational scale, used to describe the compliance of a child during induction of anesthesia. ICC contains 10 items. Score ranges from 0 to 1. 0 point indicates the behavior is not observed while 1 point means behavior is observed.
Change of parental anxiety | baseline, immediately after anesthetic induction
  The State-Trait Anxiety Inventory (STAI) is the gold standard for assessing anxiety in adults and has been used in over 1000 studies. It is comprises 20 questions. The total score ranges from 0-63. 0-9 indicates normal or no anxiety; 10-18 indicates mild to moderate anxiety; 19-29 indicates moderate to severe anxiety; and 30-63 indicates severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Olbrecht, MD, MBA, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No